CLINICAL TRIAL: NCT02854293
Title: Impact of a Booklet-Question List on Cancer Patients or Their Families Seeking Prognostic Information During a Palliative Care Consultation
Acronym: QUEPAL
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC 2011-04
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Cancer; Palliative Care
Keywords: palliative care; cancer; quality of life
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Booklet-Question List (BQL) group: 76 patients
  Interventions: Other: Booklet-Question List
- control group: Conventional palliative management
  76 patients

INTERVENTIONS:
Other: Booklet-Question List — Booklet-Question List (BQL) proposed in palliative cares, divided into 8 chapters, given to the patient before the first palliative care consultation.
  Providing a list of questions to patients and their families without any obligations allows individual adaptation of information; patients or families who are afraid of asking these questions can take advantage of this opportunity, while respecting the need to avoid these subjects for other patients
  Groups: Booklet-Question List (BQL) group

SUMMARY:
Prospective, randomized, multicentre phase III study to evaluate the level and type of information requested by patients or families during a palliative care consultation after they have been given the Booklet-Question List (BQL).

ELIGIBILITY:
Inclusion criteria:

* Patient over the age of 18 years,
* Patient who has signed the informed consent form after being given a written information sheet
* Patient followed for metastatic cancer with or without specific treatment, with a limited life expectancy
* Patient referred to the palliative care team.
* French-speaking Patient

Exclusion criteria:

* Cognitive disorders
* Documented psychiatric disorders or marked psychological fragility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient followed for metastatic cancer with or without specific treatment, with a limited life expectancy
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The number of questions asked or the concerns expressed that elicit a medical comment by the patient or the family during the palliative care consultation. | one month

SECONDARY OUTCOMES:
HADS (Hospital Anxiety and Depression Scale) anxiety and depression score | one month
QLQC-15Pal palliative quality of life score | one month
  The EORTC QLQ-C15-PAL is a questionnaire developed to assess the quality of life of palliative cancer care patients
MB coping questionnaire score | one month
  The Brief COPE is the abbreviated version of the COPE Inventory and assesses dispositional as well as situational coping efforts . The 28-item Brief COPE (consisting of 14 subscales) has acceptable psychometric properties and has been used extensively to examine the relationship between various coping strategies and psychological outcomes
Two 5-point Likert scales on information needs and satisfaction with medical information | one month
Specific questionnaire on the Booklet-Question List (mode of use, satisfaction) | one month

CONTACTS AND LOCATIONS:
Overall Officials: Carole Bouleuc, MD, Principal Investigator — Institut Curie
Locations (5):
- France (5):
  - Léon Berard, Lyon
  - Centre Alexis Vautrin, Nancy
  - Institut Curie, Paris
  - Hopital René Huguenin, Saint-Cloud
  - Polyclinique de l'Ormeau, Tarbes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouleuc C, Savignoni A, Chevrier M, Renault-Tessier E, Burnod A, Chvetzoff G, Poulain P, Copel L, Cottu P, Pierga JY, Bredart A, Dolbeault S. A Question Prompt List for Advanced Cancer Patients Promoting Advance Care Planning: A French Randomized Trial. J Pain Symptom Manage. 2021 Feb;61(2):331-341.e8. doi: 10.1016/j.jpainsymman.2020.07.026. Epub 2020 Jul 31. PMID 32739563